CLINICAL TRIAL: NCT05131321
Title: FRAME Study (Frailty-Related Ankle Fracture Management and Evaluation): Retrograde Nailing Versus Open Reduction and Internal Fixation for Unstable Fractures Around the Ankle in the Frail Elderly - A Two-Part Prospective, Randomized, Multi-Center Clinical Trial
Brief Title: FRAME Study (Frailty-Related Ankle Fracture Management and Evaluation)
Acronym: FRAME
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 119571
Record Dates: First submitted 2021-10-19; First posted 2021-11-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-03

CONDITIONS: Ankle Fractures; Pilon Fracture
Keywords: Complex ankle fracture; Pilon fracture; Primary Ankle Arthrodesis; Fragility fracture; Elderly; Open reduction; Internal fixation; AO/OTA type 44B2, B3, C1 or C2 ankle fracture
MeSH Terms: conditions — Ankle Fractures | interventions — Gene Fusion; Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Part 1: Fusion Group: Primary arthrodesis: Subjects allocated to the fusion group will have insertion of a retrograde locked calcaneal nail. Tibiotalar joint preparation, bone grafting, subtalar preparation, and fibulectomy will not be performed unless deemed necessary by the treating surgeon.
  Interventions: Procedure: Primary ankle arthrodesis (fusion)
- Part 2: Fibula: Intramedullary Fibular Nailing: Participants allocated to the IMFN group will receive a locked fibular nail using a previously described technique.
  Interventions: Procedure: Intramedullary Fibular Nailing (IMFN)
- Control Group: Internal Fixation: ORIF will be performed using modern techniques for timing and staging of fixation, soft tissue and fibula management, surgical approaches, reduction techniques, and plate choice.
  Interventions: Procedure: ORIF (open reduction and internal fixation)

INTERVENTIONS:
Procedure: Primary ankle arthrodesis (fusion) — Primary arthrodesis: Subjects allocated to the fusion group will have insertion of a retrograde locked calcaneal nail. Tibiotalar joint preparation, bone grafting, subtalar preparation, and fibulectomy will not be performed unless deemed necessary by the treating surgeon.
  Groups: Part 1: Fusion Group
Procedure: ORIF (open reduction and internal fixation) — ORIF: ORIF will be performed using modern techniques for timing and staging of fixation, soft tissue and fibula management, surgical approaches, reduction techniques, and plate choice.
  Groups: Control Group: Internal Fixation
Procedure: Intramedullary Fibular Nailing (IMFN) — Intramedullary Fibular Nailing: Participants allocated to the IMFN group will receive a locked fibular nail using a previously described technique.
  Groups: Part 2: Fibula

SUMMARY:
This will be a multi-centre randomized controlled trial, with London Health Sciences Centre (LHSC) as the lead site. Elderly patients with complex ankle fractures who meet the inclusion criteria and provide consent will be randomized (through a web-based randomization system) to one of the two treatment arms. One group (Group A) will receive primary ankle fusion, and the second group (Group B) will receive primary ankle open reduction and internal fixation (ORIF). Patient important outcomes will be compared at one year post injury

The Investigators have amended the study to include a second part for patients with less complicated but still unstable ankle fractures. In this part, patients will be randomly assigned to receive either a procedure called ORIF or another one called retrograde intramedullary fibular nailing.

DETAILED DESCRIPTION:
At the current time, there are few prospective studies comparing primary ankle arthrodesis versus Open Reduction and internal fixation (ORIF) for the treatment of complex fractures around the ankle in the frail elderly who have significant co-morbidities.

An effective alternative to ORIF that results in improved function, less post-operative pain and a lower rate of complications is desirable, particularly in the setting of a severely compromised soft tissue envelope, osteopenia or significant co-morbidities. Emerging clinical evidence regarding primary ankle fusion is encouraging, suggesting several potential benefits over ORIF in severely compromised cases including lower post-operative pain scores, improved functional outcomes, lower complication rates, and high union rates. However, high level evidence confirming these potential benefits is lacking. The results of the proposed investigation would have significant implications for the management of orthopaedic trauma patients with fragility fractures around the ankle and may in fact challenge ORIF as the gold standard of treatment in some cases.

Aims & Hypotheses

Aims:

The Investigators aim to conduct a two-part, multi-center RCT comparing retrograde nailing to ORIF for unstable fractures around the ankle in frail or compromised older adults. The primary research questions are:

Part 1: Does primary ankle fusion with a retrograde tibio-talar-calcaneal hindfoot nail for the treatment of severe fractures around the ankle (tibial pilon AO/OTA type 43 C2-3 or severe ankle fracture [fracture dislocation, severe joint impaction, severe trimalleolar) in the frail elderly result in improved outcomes and a lower rate of complications compared with ORIF?

Part 2: Does primary retrograde intramedullary fibular nailing (IMFN) result in improved outcomes compared to ORIF for frail older adults with less complex (no dislocation, no significant joint impaction), but unstable fractures(AO/OTA type 44-B2-3, C1-2) around the ankle?

Hypotheses:

The Investigators hypothesize that:

1. Retrograde nailing will result in improved health related quality of life, functional outcomes, pain and reduced complications compared to ORIF.
2. Our null hypothesis is that retrograde nailing will not result in improved post-operative health related quality of life, functional outcomes, pain, and complication rates relative to ORIF for severe fractures around the ankle in the frail elderly.

Study Design

Design:

A two-part, multi-centre randomized clinical trial (RCT)

Procedure: Patients presenting to hospital with a suspected ankle fracture will be screened and those deemed potentially eligible will be approached for consent. Consenting patients will be enrolled prospectively over a 2-year period and followed according to the research ethics board (REB) approved protocol. Patients may also consent to be contacted at 5 years to evaluate long-term changes in outcomes. Full eligibility will be determined by an orthopaedic surgeon, following appropriate radiographic scans. The local research team will measure and capture outcomes during regularly scheduled clinic or hospital visits as well as through email/phone contact for patients consenting to contact via phone/email.

ELIGIBILITY:
Patient Inclusion Criteria - Both Parts:

(i) Age ≥ 60 years (ii) One or more of the following:

* Severe soft tissue compromise
* Significant co-morbidities (vascular disease + chronic trophic changes, diabetes + neuropathy, chronic renal failure, morbid obesity (BMI> 40))
* Frailty as defined by a Dalhousie Clinical Frailty Scale score ≥4

Part 1 Specific Inclusion Criteria:

(i) Isolated fracture (within 4 weeks of injury): an AO/OTA type 43C2 or C3 tibial pilon fracture or severe ankle fracture (fracture-dislocation, severe joint impaction, severe trimalleolar)

Part 2 Specific Inclusion Criteria (i) Isolated fracture (within 4 weeks of injury): an AO/OTA type 44B2, B3, C1 or C2 ankle fracture

Patient Exclusion Criteria - Both Parts:

(i) Presence of vascular injury or pathologic fracture; (ii) Previous tibia pilon fracture or retained hardware in affected limb; (iii) Refusal to participate; (iv) Inability to obtain informed consent due to language barrier

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ankle fracture patients receiving care at the participating institutions will be eligible for enrolment based on the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Short-Form 12 (SF-12). | 1 year post-surgery.
  • The primary outcome will be health related quality of life, measured by the SF-12 at one year post surgery. The SF12 measures patient reported, health related quality of life from 0 to 100, with higher scores indicating better physical and mental health functioning.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | 1 year post-surgery
  • Pain will be measured on a scale of 0 to 10 with 0 being no pain and 10 being the worst pain imaginable.
Function IndeX (FIX-IT) | 1 year post-surgery
  • Weight-bearing will be assessed by the FIX-IT score, which provides a simple, standardized and validated approach to assess weight bearing and pain from 0 to 12 with 12 being no pain or weigh-bearing limitations.
Euro-Qol-5 Dimension (EQ5D) | 1 year post-surgery
  • Health-related quality of life will also be measured by the EQ5D. The EQ5D measures patient-reported health related quality of life from 0 to 100, with 100 being the best health imaginable.
PROMIS-Physical Function Short Form (PROMIS-PF), version 10a | 1 year post-surgery
  • Patient-reported function will be measured via the PROMIS-PF Short form, a rigorously developed, patient-centred measure that measures functional ability from 10 to 50, with 50 being no functional limitations.
Olerud Molander Ankle Score (OMAS) | 1 year post-surgery
  • Patient-reported, ankle fracture specific functional ability will be measured by the OMAS. The OMAS is scored from 0 to 100 with higher scorings representing better functional ability.
Extended Timed-up and Go (TUG) Test | 1 year post-surgery
  • Patient mobility will be measured by the Extended TUG test. To ensure that the investigators remain unbiased during the evaluation and follow-up process, the TUG test will be administered by independent assessors blinded to treatment allocation. The TUG test record the amount of time a patient requires to stand from a chair, walk 3 metres, turn and walk back to sit on the chair. The patient is allowed to use their regular walking aids, and the use of walking aids is recorded by the assessor. A shorter time represents better patient mobility.
Rate of complications | 1 year post-surgery
  • The rate of complications, including nonunion, malunion, infection, implant failure, arthritis, and re-operation will be captured.
Foot and Ankle Ability Measure (FAAM) | [Time Frame: 1 year post-surgery]
  • Patient-reported, ankle fracture specific functional ability will be measured by the OMAS. The OMAS is scored from 0 to 100 with higher scorings representing better functional ability.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided